CLINICAL TRIAL: NCT04374487
Title: A Phase II, Open Label, Randomized Controlled Trial to Assess the Safety and Efficacy of Convalescent Plasma to Limit COVID-19 Associated Complications
Brief Title: Assess the Safety and Efficacy of Convalescent Plasma to Limit COVID-19 Associated Complications
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Max Healthcare Insititute Limited (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MHC-COVID-19-CP
Record Dates: First submitted 2020-04-29; First posted 2020-05-05 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: COVID 19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Arm (Experimental): 50 subjects will be randomized in this arm. Patients in the test group will receive convalescent plasma.
  Interventions: Drug: Convalescent Plasma
- Control Arm (Other): 50 subjects will be randomized in this arm and will be treated according to the standard care. The Ministry of Health and Welfare has issued detailed guidelines for the management of sCOVID-19 based on varying grades of severity. For the management of ARDS or sepsis, the respective guidelines issued by ARDSNet and Surviving Sepsis campaign will be followed. Other institutional protocols for supportive management will be implemented.
  Interventions: Other: Standard Care Therapy

INTERVENTIONS:
Drug: Convalescent Plasma — 200 ml of ABO compatible plasma transfusion will be done to the subject randomized for the test arm therapy
  Arms: Test Arm
Other: Standard Care Therapy — Subjects randomized to control group will be on standard care treatment according to Institutional Protocols.
  Arms: Control Arm

SUMMARY:
The novel coronavirus disease (COVID-19), which began in Wuhan, China, in December 2019, has been declared to be a pandemic by the World Health Organization (WHO), Caused by the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), COVID-19 has resulted in 1,781,127 cases and 108,994 deaths globally (till 12th April, 2020), affecting 199 countries and 2 international conveyances. US FDA has recently approved Convalescent Plasma from patients recovered from COVID 19 for the treatment of severe or life threatening COVID-19 infections. In a small case series, five critically ill COVID-19 patients with ARDS were treated with convalescent plasma containing neutralizing antibodies. Infusion of plasma was followed by improvement in clinical status in all five patients, with no deaths and the study reported that three patients were discharged, whilst two continued to be stable on mechanical ventilation. We designed this phase II, open label, randomized clinical trial with the primary objective to assess the safety and efficacy of the therapy in the second stage.

DETAILED DESCRIPTION:
The study will be conducted over the period of one year on 100 Hospitalized, COVID-19 patients, fulfill the inclusion and exclusion criteria, and are admitted for care at COVID-19 management facilities in Max healthcare Hospital will be eligible for inclusion in the trial. This Phase II, open label, randomized controlled trial. Consecutive patients meeting the inclusion-exclusion criteria and providing informed consent will be randomly assigned to the test and the control group using random numbers generated by randomization.com. Patients in the test group will receive convalescent plasma and the control group will be on standard care.

COVID-19 convalescent plasma will be collected from recovered individuals if they are eligible to donate blood. For infusion of plasma existing SOP of the wards w.r.t transfusion of FFP should be followed with special care to monitor these patients during and post-24 hours of transfusion. An ABO compatible plasma bag of approx. 200ml will be issued maintaining all the blood bank records after thawing at 37 degree Celsius. The first plasma transfusion may be followed by one or two additional doses of 200 ml at 24 hours interval according to disease severity and tolerance of the infusions. Baseline data about the demography, clinical presentations, ongoing medical therapy, and clinical history of participants in both arms will be collected and compared. Response to convalescent plasma will be coded as a binary outcome - based on whether the composite primary end point is met or not. Adverse events associated with infusion of convalescent plasma will also be descriptively summarized and compared with the adverse events experienced by participants receiving standard of care.

Eligibility of Potential Donor

1. Only males and nulliparous female donors of weight > 55 kgs will be included.
2. Donor eligibility criteria for whole blood donation as per the departmental SOP will be followed in accordance to the Drugs & Cosmetics Act 1940 and rules 1945 therein (as amended till March 2020). Donor will be screened, followed by brief physical examination.
3. Donors not fit to donate blood based on the history and examination will be deferred and excluded from plasma donor pool for a time period specified by country regulation & departmental SOPs.
4. In addition to the aforementioned donor eligibility criteria, two EDTA samples (5 ml each) and one plain sample (5 ml) will be drawn for the following pre-donation tests as required for convalescent plasmapheresis (CPP).

   * Blood group and antibody screening - Antibody screen positive donors will be deferred.
   * Complete blood count including Hb, Hct, Platelet count, Total and differential leucocyte count. Donors with Hb>12.5g/dl, platelet count >1, 50,000 per microliter of blood and TLC within normal limits will be accepted.
   * Screening for HIV, HBV and HCV by serology and NAT. Donor negative by both the tests will be included.
   * Screening for syphilis and malaria by serology. Negative donors will be included
   * Total serum protein. Donors with total serum protein > 6gm/dl will be accepted (as per Drugs and Cosmetics (Second Amendment) Rules, 2020)
   * Titration of anti-COVID-19 (both IgG and IgM) antibodies and SARS- CoV-2 neutralizing antibodies may be done depending on availability of facilities at the time of testing. (Desired titers for IgG antibodies >1024 or neutralizing antibodies >40) doubling dilution of donor serum will be done and titration will be done using ELISA. If not done at the time of plasma collection the donor samples will be stored in aliquots at <-80° C to be tested at a later date.
   * Molecular test for COVID-19 either from nasopharyngeal swab specimens or blood may be done depending on availability of tests. Donors positive will be deferred.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients admitted with RT-PCR confirmed COVID-19 illness. 2. Age > 18 years 3. Written informed consent 4. Has any of the two

  1. PaO2/ FiO2 <300
  2. Respiratory Rate > 24/min and SaO2 < 93% on room air

Or In case of Severe or immediately life-threatening COVID-19, for example:

a. Severe disease is defined as: i. dyspnea, ii. respiratory frequency ≥ 30/min, iii. blood oxygen saturation ≤ 93%, iv. partial pressure of arterial oxygen to fraction of inspired oxygen ratio < 300, and/or v. lung infiltrates > 50% within 24 to 48 hours b. Life-threatening disease is defined as: i. respiratory failure, ii. septic shock, and/or iii. multiple organ dysfunction or failure

Exclusion Criteria:

* 1. Pregnant women 2. Breastfeeding women 3. Known hypersensitivity to blood products 4. Receipt of Pooled Immunoglobulin in last 30 days 5. Participating in any other clinical trial 6. Clinical status precluding infusion of blood products

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-05-09 (Actual); Primary Completion 2021-08-09 (Estimated); Study Completion 2021-08-09 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is a composite measure of the avoidance of - 1. Progression to severe ARDS (P/F ratio 100) and 2. All-cause Mortality at 28 days | depends on the total treatment time of the subjects within one year period of the trial.
  Baseline data about the demography, clinical presentations, ongoing medical therapy, and clinical history of participants in both arms will be collected and compared. Response to convalescent plasma will be coded as a binary outcome - based on whether the composite primary end point is met or not. All the statistical tests will be done at 5% level of significance and SPSS21 will be used for calculations.

SECONDARY OUTCOMES:
Time to symptom resolution-Fever,Shortness of Breath,Fatigue | one year
  Data from both arm will be collected and compared time to time
Hospital length of stay | one year
  total time of stay at hospital for the treatment and cure will be calculated and compared of both the arms
Change in SOFA pre and post transfusion | one year
  sepsis-related organ failure assessment (SOFA) score will be calculated for both the arms and compared for the analysis.
Duration of respiratory support required a. Duration of Invasive Mechanical Ventilation b. Duration of Non-Invasive | one year
  Most COVID patients admitted to intensive care require some form of respiratory support. Whether or not the plasma therapy decreases the duration of respiratory support and its comparison with the standard care therapy will be calculated.
Radiological improvement | one year
  Comparison between group response rates will be analyzed by radiological imaging and reported.
Adverse events (AE) associated with transfusion | one year
  Adverse events associated with infusion of convalescent plasma will also be descriptively summarized and compared with the adverse events experienced by participants receiving standard of care.
To measure the change in RNA levels (Ct values) of SARS-CoV-2 from RT-PCR [Time Frame: Days 0, 1, 3, and 7 after transfusion] | one year
  Ct values from day 0, 1, 3 & 7 will be calculated by RT-PCR and compared to check the response of therapy on the viral load. All the statistical tests will be done at 5% level of significance and SPSS21 will be used for calculations.
Levels of bio-markers pre and post transfusion | one year
  Bio-markers can play a role in understanding how existing drugs can be used to treat Covid-19. Hence, pre and post Plasma transfusion the level of bio-markers will be checked and compared.
Need of Vasopressor use | one year
  For critically ill subjects in both the arms the need of vasopressor will be compared. All these comparisons are for qualitative data and will be assessed for statistical significance by Fisher exact test in view of the small sample size.

CONTACTS AND LOCATIONS:
Overall Officials: Sangeeta Pathak, MBBS,Diploma, Principal Investigator — Max Super Speciality Hospital, Saket (DDF)
Locations (1):
- Max Super Speciality hospital, Saket (A unit of Devki Devi Foundation), New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No